CLINICAL TRIAL: NCT04148846
Title: COMPARATION BETWEEN SPHENOPALATINE BLOCK AND MULTIMODAL CLINICAL TREATMENT IN TREATMENT OF HEADACHE AFTER DURAL PUNCTION IN PREGNANT WOMEN.
Brief Title: Sphenopalatine Blockade Versus Clinical Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06860018.0.0000.0068
Record Dates: First submitted 2019-10-30; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-09

CONDITIONS: Headache, Post-Dural Puncture
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Sphenopalatine Ganglion Block; Ketoprofen; Gabapentin; Dexamethasone; Theophylline

STUDY DESIGN:
Intervention Model Description: A prospective randomized clinical, analytical study will be conducted at the Obstetric Center of the Central Institute of the University of São Paulo School of Medicine Clinical Hospital (ICHC-FMUSP). Postpartum women undergoing neuraxial block for cesarean section, vaginal delivery or uterine curettage, and who later present with cerebrospinal fluid hypotension, will be studied after evaluation and diagnosis by anesthesiologist. The research will be submitted for evaluation by the Research Ethics Committees, according to resolution 196/96. Patients will be approached as to the eligibility of their participation in the study, and after the necessary clarifications, will authorize or not the proposed interventions and data collection, by signing the Informed Consent Form.
Who Masked: Participant
Masking Description: The patients will be randomly divided into three groups according to the reduced distribution of use of the site www.randomization.com to be conducted prior to the commencement of surveys and data collection. Each patient is given an identification number following a search entry order, and this number is already available through prior randomization linked to one of the three intervention groups. The professional who administers as drugs will be external to the research group and may cause non-burdensome form. Researchers who perform the evaluations of the researched variables can obtain the following results for the intervention performed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clinical treatment - old protocol (Active Comparator): In group I, patients will receive clinical treatment according to the institution's old protocol for post dural puncture headache.
  Interventions: Drug: Dypirone; Drug: Ketoprofen
- Clinical treatment - new protocol (Active Comparator): In group II, patients will receive clinical treatment, according to the new protocol of the institution.
  Interventions: Drug: Dypirone; Drug: Ketoprofen; Drug: Gabapentin; Drug: Dexamethasone; Drug: Theophylline; Dietary Supplement: Espresso coffee
- Sphenopalatine block (Experimental): In group III patients will receive clinical treatment, according to the new protocol of the institution, associated with sphenopalatine block.
  Interventions: Drug: Dypirone; Procedure: Sphenopalatine block; Drug: Ketoprofen; Drug: Gabapentin; Drug: Dexamethasone; Drug: Theophylline; Dietary Supplement: Espresso coffee

INTERVENTIONS:
Drug: Dypirone — Dipyrone 2g, 6 / 6h for 7 days, orally or intravenous
Procedure: Sphenopalatine block — The sphenopalatine block will be performed with the patient in the supine position, with neck extended. Following topical anesthesia of the nasal vestibules with one application of 10% lidocaine spray and one application of 2% lidocaine gel in each nostril, two long cotton swab applicators embedded in 2% lidocaine jelly, one in each nostril, will be introduced. They will be advanced at a 45-degree angle to the floor of the nose until resistance is encountered, indicating that the swab is in the posterior nasopharyngeal wall, superior to the middle nasal concha. It will be held in this position for 5 minutes and then removed. Thereafter, a 14 gauge, non-cutting, teflon blunt catheter will be introduced into each nostril at a 45 ° angle to the hard palate until it touches the posterior wall of the nasopharynx. For it will be applied 2ml of 0.375% Ropivacaine, on each side, slowly.
  Arms: Sphenopalatine block
Drug: Ketoprofen — Ketoprofen 100 mg, 12 / 12h for 5 days, orally or intravenous
Drug: Gabapentin — Gabapentin 300 mg 8 / 8h for 7 days orally
  Arms: Clinical treatment - new protocol; Sphenopalatine block
Drug: Dexamethasone — Dexamethasone 4mg 8 / 8h for 48h orally
  Arms: Clinical treatment - new protocol; Sphenopalatine block
Drug: Theophylline — Theophylline 200mg, 12 / 12h, for 5 days, orally
  Arms: Clinical treatment - new protocol; Sphenopalatine block
Dietary Supplement: Espresso coffee — Espresso coffee 20ml, 5x / day, for 7 days
  Arms: Clinical treatment - new protocol; Sphenopalatine block

SUMMARY:
Post-dural puncture headache leads to high morbidity and cost to the health system. Pregnant women have a higher incidence than other population groups. There are several treatments for post dural puncture headache mentioned in the literature, not all well established, with a wide heterogeneity of treatment between services. Sphenopalatine block then appears as an alternative treatment, having been described as effective in reports and case series, requiring comparative experimental studies.

DETAILED DESCRIPTION:
Post-dural puncture headache leads to high morbidity and cost to the health system. Pregnant women have a higher incidence than other population groups. There are several treatments for post dural puncture headache mentioned in the literature, not all well established, with a wide heterogeneity of treatment between services. Sphenopalatine block then appears as an alternative treatment, having been described as effective in reports and case series, requiring comparative experimental studies.

OBJECTIVES: To evaluate the efficacy of sphenopalatine blockade in combination with multimodal treatment in reducing the incidence of epidural blood patch and pain intensity in patients who develop headache after dural puncture, compared with the clinical treatment in our service.

METHODS: A prospective randomized clinical, analytical study will be conducted at the Obstetric Center of the Central Institute of the University of São Paulo School of Medicine Hospital das Clínicas (ICHC-FMUSP). Women will be included who will undergo neuroaxis block for cesarean section, vaginal delivery or uterine curettage, and who later present headache after dural puncture, after evaluation and diagnosis by anesthesiologist. The patients will be divided into three groups at random. In group I, patients will receive clinical treatment according to the institution's old protocol for post dural puncture headache. In group II, patients will receive clinical treatment, according to the new protocol of the institution. In group III patients will receive clinical treatment, according to the new protocol of the institution, associated with sphenopalatine block. They will be reevaluated after 12, 24 and 48 hours, and a visual analog scale will be applied to evaluate improvement. The pain will be quantified before and after treatment. Pain intensity will be evaluated by verbal numerical scale (EVN), incidence of need for epidural blood buffer in each group, as well as length of hospital stay (in days).

ELIGIBILITY:
Inclusion Criteria:

* women who will undergo neuroaxis block for cesarean section, vaginal delivery or uterine curettage, and who later present with cerebrospinal fluid hypotension headache, after evaluation and diagnosis by anesthesiologist.

Exclusion Criteria:

* patients previously diagnosed with chronic headache; patients with contraindication for neuraxial anesthesia, patients with contraindication for any drugs involved in the study and users of psychotropic intravenous drugs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-09-25 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
Pain scores | 2 days
  Headache intensity will be assessed using a numerical verbal scale (EVN) from 0 to 10, with 0 being no pain and 10 being the worst possible pain. Patients will quantify pain before and after treatment. Will be reevaluated after 12, 24 and 48 hours.

SECONDARY OUTCOMES:
Satisfaction with treatment | 2 days
  Satisfaction with pain management will be assessed using a numerical scale from 0 to 10, with 0 being unsatisfied and 10 being complete satisfaction. Will be reevaluated after 12, 24 and 48 hours.
Basic newborn care | 2 days
  At each moment of evaluation, patients will be asked about any difficulty in breastfeeding or performing basic newborn care.
Blood patch incidence | 2 days
  The incidence of blood patch in each group will be quantified if necessary.
Length of hospital stay | 2 days
  Evaluate how long hospital stay of each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Hermann S Fernandes, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No